CLINICAL TRIAL: NCT01869088
Title: Phase Ⅲ Trial of Transcatheter Arterial Chemoembolization(TACE) Plus Recombinant Human Adenovirus Type 5 Injection for Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: TACE Plus Recombinant Human Adenovirus for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-120402
Record Dates: First submitted 2013-02-16; First posted 2013-06-05 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE; Carcinoma,Hepatocellular; Liver Neoplasms; overall survival; Recombinant Human Adenovirus Type 5 Injection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE Only (Active Comparator): TACE with chemothrapy drugs (E-ADM 50mg, Lobaplatin 50 mg, MMC 6mg)and followed with embolization with lipiodol or/and polyvinyl alcohol particles.
  Interventions: Procedure: Transartery Chemoembolization
- TACE Plus Adenovirus (Experimental): After identifying the target artery of HCC, Recombinant Human Adenovirus Type 5 Injection（15.0*1011vp：0.5ml*3） will be first infused through the target artery of HCC patient and followed with chemothrapy drugs (E-ADM 50mg, Lobaplatin 50 mg, MMC 6mg) and lipiodol emulsion or/and polyvinyl alcohol particles(dependent on the tumor size) Procedure: TACE (Transcatheter arterial chemoembolization)
  Interventions: Drug: Recombinant Human Adenovirus Type 5 Injection; Procedure: Transartery Chemoembolization

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 Injection — After identifying the target artery of HCC, Recombinant Human Adenovirus Type 5 Injection（15.0*1011vp：0.5ml*3） will be first infused through the target artery
  Arms: TACE Plus Adenovirus
Procedure: Transartery Chemoembolization — Transartery chemoembolization with chemothrapy drugs (E-ADM 50mg, Lobaplatin 50 mg, MMC 6mg)and followed with embolization with lipiodol or/and polyvinyl alcohol particles.

SUMMARY:
The purpose of this study is to determine if TACE plus Recombinant Human Adenovirus Type 5 Injection will improve outcome in patients with advanced hepatocellular carcinoma (HCC) not amenable to surgery or local ablative therapy.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is currently one of the mainstays of palliative treatments worldwide for patients with unresectable Hepatocellular Carcinoma(HCC).However, the long term outcomes were generally poor for HCC patients treated with TACE. Recombinant Human Adenovirus Type 5, an E1B gene deleted adenovirus, is known to have a significant antitumor activity. In addition, local injection of recombinant human adenovirus type 5 can enhance the effect of antitumor therapies (chemotherapy and radiotherapy). The hypothesis is that patients with unresectable HCC may benefit from recombinant human adenovirus type 5 in combination with TACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed as HCC according to European Association for Study of the Liver criteria.
* BCLC stage A or B
* Child-Pugh class A or B (Child-Pugh score 7)
* ECOG performance status of 0
* Patients must have at least one tumor lesion that meets both of the following criteria:

  * The lesion can be accurately measured in at least one dimension according to RECIST criteria
  * The lesion has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
  * Patients who have received previous local therapy treatments (RFA, PEI, cryoablation, surgery, resection) to non-target lesions are eligible
  * Local therapy must have been completed at least 4 weeks prior to baseline scan.
* Haematology:Absolute neutrophil count (ANC) > 1 x 109/L, Platelet count > 40 x 109/L, Haemoglobin > 9 g/dL (may be transfused to maintain or exceed this level) Prothrombin time international normalized ratio < 1.5
* Biochemistry:Total bilirubin < 2 mg/dL Serum creatinine < 1.5 x the upper limit of normal
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Tumor factors

  * Presence of extrahepatic metastasis
  * Predominantly infiltrative lesion
  * Diffuse tumor morphology with extensive lesions involving both lobes.
* Vascular complications

  * Hepatic artery thrombosis, or
  * Partial or complete thrombosis of the main portal vein, or
  * Tumor invasion of portal branch of contralateral lobe, or
  * Hepatic vein tumor thrombus, or
  * Significant arterioportal shunt not amenable to shunt blockage
* Liver function

  * Advanced liver disease: ascites, hepatic encephalopathy
  * Patients with clinically significant gastrointestinal bleeding within the 30 days prior to study entry.
* Others

  * Renal failure requiring hemo- or peritoneal dialysis
  * Pregnant or lactating women.
  * Active sepsis or bleeding.
  * Hypersensitivity to intravenous contrast agents.
  * The patient has received prior treatment for HCC target lesion.
  * History of cardiac disease

    * Congestive heart failure > NYHA class 2; active coronary artery disease
    * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management.
  * Serious non-healing wounds (including wounds healing by secondary intention), acute or non-healing ulcers, or bone fractures within 3 months.
  * The patient is, in the opinion of the investigator, unable and / or unwilling to comply with treatment and study instructions.
  * Substance abuse (current), psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
  * Any active clinically serious infections (> grade 2 NCI-CTCAE ver 3.0)
  * HIV infection or AIDS-related illness or serious acute or chronic illness (based on medical history)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | 3 years

SECONDARY OUTCOMES:
Number of adverse events | 30 days
  Number of adverse events, and number of patients who developed adverse event. Postoperative adverse events were graded based on the Common Terminology Criteria for Adverse Events ( CTCAE )
Tumor response | 12 weeks
  Tumor response based on modified RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Vogl TJ, Trapp M, Schroeder H, Mack M, Schuster A, Schmitt J, Neuhaus P, Felix R. Transarterial chemoembolization for hepatocellular carcinoma: volumetric and morphologic CT criteria for assessment of prognosis and therapeutic success-results from a liver transplantation center. Radiology. 2000 Feb;214(2):349-57. doi: 10.1148/radiology.214.2.r00fe06349. PMID 10671580
- [Result] Ono Y, Yoshimasu T, Ashikaga R, Inoue M, Shindou H, Fuji K, Araki Y, Nishimura Y. Long-term results of lipiodol-transcatheter arterial embolization with cisplatin or doxorubicin for unresectable hepatocellular carcinoma. Am J Clin Oncol. 2000 Dec;23(6):564-8. doi: 10.1097/00000421-200012000-00006. PMID 11202797
- [Result] Geschwind JF, Ramsey DE, Cleffken B, van der Wal BC, Kobeiter H, Juluru K, Hartnell GG, Choti MA. Transcatheter arterial chemoembolization of liver tumors: effects of embolization protocol on injectable volume of chemotherapy and subsequent arterial patency. Cardiovasc Intervent Radiol. 2003 Mar-Apr;26(2):111-7. doi: 10.1007/s00270-002-2524-6. Epub 2003 Mar 6. PMID 12616414
- [Result] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Bruix J, Llovet JM, Castells A, Montana X, Bru C, Ayuso MC, Vilana R, Rodes J. Transarterial embolization versus symptomatic treatment in patients with advanced hepatocellular carcinoma: results of a randomized, controlled trial in a single institution. Hepatology. 1998 Jun;27(6):1578-83. doi: 10.1002/hep.510270617. PMID 9620330
- [Result] Camma C, Schepis F, Orlando A, Albanese M, Shahied L, Trevisani F, Andreone P, Craxi A, Cottone M. Transarterial chemoembolization for unresectable hepatocellular carcinoma: meta-analysis of randomized controlled trials. Radiology. 2002 Jul;224(1):47-54. doi: 10.1148/radiol.2241011262. PMID 12091661
- [Result] Lee KH, Liapi E, Vossen JA, Buijs M, Ventura VP, Georgiades C, Hong K, Kamel I, Torbenson MS, Geschwind JF. Distribution of iron oxide-containing Embosphere particles after transcatheter arterial embolization in an animal model of liver cancer: evaluation with MR imaging and implication for therapy. J Vasc Interv Radiol. 2008 Oct;19(10):1490-6. doi: 10.1016/j.jvir.2008.06.008. Epub 2008 Aug 27. PMID 18755602
- [Result] Higashi S, Tabata N, Kondo KH, Maeda Y, Shimizu M, Nakashima T, Setoguchi T. Size of lipid microdroplets effects results of hepatic arterial chemotherapy with an anticancer agent in water-in-oil-in-water emulsion to hepatocellular carcinoma. J Pharmacol Exp Ther. 1999 May;289(2):816-9. PMID 10215657
- [Result] Caturelli E, Siena DA, Fusilli S, Villani MR, Schiavone G, Nardella M, Balzano S, Florio F. Transcatheter arterial chemoembolization for hepatocellular carcinoma in patients with cirrhosis: evaluation of damage to nontumorous liver tissue-long-term prospective study. Radiology. 2000 Apr;215(1):123-8. doi: 10.1148/radiology.215.1.r00ap21123. PMID 10751477
- [Result] Llovet JM, Bustamante J, Castells A, Vilana R, Ayuso Mdel C, Sala M, Bru C, Rodes J, Bruix J. Natural history of untreated nonsurgical hepatocellular carcinoma: rationale for the design and evaluation of therapeutic trials. Hepatology. 1999 Jan;29(1):62-7. doi: 10.1002/hep.510290145. PMID 9862851
- [Result] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Result] Lau WY, Yu SC, Lai EC, Leung TW. Transarterial chemoembolization for hepatocellular carcinoma. J Am Coll Surg. 2006 Jan;202(1):155-68. doi: 10.1016/j.jamcollsurg.2005.06.263. Epub 2005 Oct 19. No abstract available. PMID 16377509
- [Result] Lee KH, Liapi E, Ventura VP, Buijs M, Vossen JA, Vali M, Geschwind JF. Evaluation of different calibrated spherical polyvinyl alcohol microspheres in transcatheter arterial chemoembolization: VX2 tumor model in rabbit liver. J Vasc Interv Radiol. 2008 Jul;19(7):1065-9. doi: 10.1016/j.jvir.2008.02.023. Epub 2008 Apr 10. PMID 18589321
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Groupe d'Etude et de Traitement du Carcinome Hepatocellulaire. A comparison of lipiodol chemoembolization and conservative treatment for unresectable hepatocellular carcinoma. N Engl J Med. 1995 May 11;332(19):1256-61. doi: 10.1056/NEJM199505113321903. PMID 7708069
- [Result] Yoon JH, Kim HC, Chung JW, Yoon JH, Jae HJ, Park JH. CT findings of completely regressed hepatocellular carcinoma with main portal vein tumor thrombosis after transcatheter arterial chemoembolization. Korean J Radiol. 2010 Jan-Feb;11(1):69-74. doi: 10.3348/kjr.2010.11.1.69. Epub 2009 Dec 28. PMID 20046497
- [Result] Rieger R, Whitacre D, Cantwell MJ, Prussak C, Kipps TJ. Chimeric form of tumor necrosis factor-alpha has enhanced surface expression and antitumor activity. Cancer Gene Ther. 2009 Jan;16(1):53-64. doi: 10.1038/cgt.2008.57. Epub 2008 Jul 25. PMID 18654609
- [Result] Shi M, Wang F, Liu M, Zhang B, Qiu Z, Lei Z, Masayoshi N, Gao L, Wu Z. [Adenovirus-mediated transfer of human wild-type p53, GM-CSF, and B7-1 genes efficiently produces growth suppression and apoptosis of hepatocellular cells in vitro]. Zhonghua Gan Zang Bing Za Zhi. 2001 Aug;9(4):229-31. Chinese. PMID 11602056
- [Result] Shi M, Wang FS, Wu ZZ. Synergetic anticancer effect of combined quercetin and recombinant adenoviral vector expressing human wild-type p53, GM-CSF and B7-1 genes on hepatocellular carcinoma cells in vitro. World J Gastroenterol. 2003 Jan;9(1):73-8. doi: 10.3748/wjg.v9.i1.73. PMID 12508355
- [Result] Guo Y, Zeng Y, Wang K, Zhu X, Luo H, Zheng M, Li M, Chen J. [Therapeutic potential of recombinant adenovirus expressing p53 in hepatocellular carcinoma cell lines]. Zhonghua Gan Zang Bing Za Zhi. 2001 Jul;9 Suppl:43-5. Chinese. PMID 11509137
- [Result] He Q, Liu Y, Zou Q, Guan YS. Transarterial injection of H101 in combination with chemoembolization overcomes recurrent hepatocellular carcinoma. World J Gastroenterol. 2011 May 14;17(18):2353-5. doi: 10.3748/wjg.v17.i18.2353. PMID 21633603
- [Result] Choi JY, Park YM, Byun BH, Kim BS, Hong EG, Shin DY, Seong YR, Im DS. Adenovirus-mediated p53 tumor suppressor gene therapy against subcutaneous HuH7 hepatoma cell line nodule of nude mice. J Korean Med Sci. 1999 Jun;14(3):271-6. doi: 10.3346/jkms.1999.14.3.271. PMID 10402169
- [Result] Chen CA, Lo CK, Lin BL, Sibley E, Tang SC. Application of doxorubicin-induced rAAV2-p53 gene delivery in combined chemotherapy and gene therapy for hepatocellular carcinoma. Cancer Biol Ther. 2008 Feb;7(2):303-9. doi: 10.4161/cbt.7.2.5333. Epub 2007 Nov 21. PMID 18059187
- [Result] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Result] Mullen JT, Tanabe KK. Viral oncolysis. Oncologist. 2002;7(2):106-19. doi: 10.1634/theoncologist.7-2-106. PMID 11961194
- [Result] Benedict CA, Norris PS, Prigozy TI, Bodmer JL, Mahr JA, Garnett CT, Martinon F, Tschopp J, Gooding LR, Ware CF. Three adenovirus E3 proteins cooperate to evade apoptosis by tumor necrosis factor-related apoptosis-inducing ligand receptor-1 and -2. J Biol Chem. 2001 Feb 2;276(5):3270-8. doi: 10.1074/jbc.M008218200. Epub 2000 Oct 24. PMID 11050095
- [Result] Hamid O, Varterasian ML, Wadler S, Hecht JR, Benson A 3rd, Galanis E, Uprichard M, Omer C, Bycott P, Hackman RC, Shields AF. Phase II trial of intravenous CI-1042 in patients with metastatic colorectal cancer. J Clin Oncol. 2003 Apr 15;21(8):1498-504. doi: 10.1200/JCO.2003.09.114. PMID 12697873
- [Result] Bauzon M, Castro D, Karr M, Hawkins LK, Hermiston TW. Multigene expression from a replicating adenovirus using native viral promoters. Mol Ther. 2003 Apr;7(4):526-34. doi: 10.1016/s1525-0016(03)00023-6. PMID 12727116
- [Result] Hermiston TW, Kuhn I. Armed therapeutic viruses: strategies and challenges to arming oncolytic viruses with therapeutic genes. Cancer Gene Ther. 2002 Dec;9(12):1022-35. doi: 10.1038/sj.cgt.7700542. PMID 12522441
- [Result] Khuri FR, Nemunaitis J, Ganly I, Arseneau J, Tannock IF, Romel L, Gore M, Ironside J, MacDougall RH, Heise C, Randlev B, Gillenwater AM, Bruso P, Kaye SB, Hong WK, Kirn DH. a controlled trial of intratumoral ONYX-015, a selectively-replicating adenovirus, in combination with cisplatin and 5-fluorouracil in patients with recurrent head and neck cancer. Nat Med. 2000 Aug;6(8):879-85. doi: 10.1038/78638. PMID 10932224
- [Result] Nemunaitis J, Khuri F, Ganly I, Arseneau J, Posner M, Vokes E, Kuhn J, McCarty T, Landers S, Blackburn A, Romel L, Randlev B, Kaye S, Kirn D. Phase II trial of intratumoral administration of ONYX-015, a replication-selective adenovirus, in patients with refractory head and neck cancer. J Clin Oncol. 2001 Jan 15;19(2):289-98. doi: 10.1200/JCO.2001.19.2.289. PMID 11208818
- [Result] Kirn D. Oncolytic virotherapy for cancer with the adenovirus dl1520 (Onyx-015): results of phase I and II trials. Expert Opin Biol Ther. 2001 May;1(3):525-38. doi: 10.1517/14712598.1.3.525. PMID 11727523